CLINICAL TRIAL: NCT06741072
Title: A Phase 1B Double Blinded Randomized Trial Evaluating Safety, Tolerability, and Immune Response of OSU-2131 a BZLF1 Peptide Vaccine With Stimulon™ QS-21 Solution Adjuvant in Healthy Volunteers and Patients Awaiting Solid Organ Transplantation
Brief Title: BZLF1 Peptide Vaccine (OSU-2131) With QS-21 for the Prevention of Epstein-Barr Virus Related Cancer in Patients Awaiting Solid Organ Transplants
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: study drug issue
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Timothy Voorhees, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-20219; NCI-2024-09778 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease, Stage 4; Chronic Kidney Disease, Stage 5; EBV-Related Lymphoproliferative Disorder; EBV-Related Malignant Neoplasm; Post-Transplant Lymphoproliferative Disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Specimen Handling; Protein Subunit Vaccines; saponin QA-21V1; Quillaja Saponins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Healthy volunteers, patients, and site staff evaluating the patients will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (OSU-2131, QS-21) (Experimental): Healthy volunteers and patients receive OSU-2131 SC with QS-21 SC on day 0, and weeks 2 and 4 in the absence of unacceptable toxicity or patient proceeds to transplant. Healthy volunteers and patients additionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Peptide Vaccine; Biological: QS21
- Group II (placebo) (Placebo Comparator): Healthy volunteers receive PBS SC on day 0, and weeks 2 and 4 in the absence of unacceptable toxicity. Healthy volunteers additionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Dulbecco''s Phosphate-Buffered Saline

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Dulbecco''s Phosphate-Buffered Saline — Given SC
  Other Names: DPBS; PBS; Phosphate-Buffered Saline
  Arms: Group II (placebo)
Biological: Peptide Vaccine — Given OSU-2131 SC
  Arms: Group I (OSU-2131, QS-21)
Biological: QS21 — Given SC
  Other Names: NIAID VEU 016; Purified Quillaja Saponin; QS-21; QS-21 Adjuvant; QUILLAJA SAPONIN (QS-21); Stimulon QS-21 Adjuvant
  Arms: Group I (OSU-2131, QS-21)

SUMMARY:
This phase 1B trial tests the safety, side effects and best dose of rh-Hsc70- BZLF1 peptide complex (OSU-2131) with Stimulon (Trademark) QS-21 and evaluates how well it works in preventing Epstein-Barr virus (EBV) infection and related cancers in healthy volunteers and patients awaiting a solid organ transplant. Currently, patients who receive an organ transplant receive immune suppression therapy which can make it harder for the body to fight infections. This treatment also increases the risk for cancers that are triggered by the EBV. Vaccines made from synthetic peptide (RAKFKQLL) derived from the BZLF1 protein, may help the body build an effective immune response against EBV infections. QS-21, a saponin adjuvant, is a substance from plants that, when given with vaccine therapy, may improve the way the immune system responds to disease. Giving OSU-2131 with QS-21 may help the immune system fight EBV and protect against EBV infection and the cancers that it can cause in patients awaiting solid organ transplants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the overall safety profile of three different dose levels of OSU-2131 vaccination each with 50 mcg Stimulon (Trademark) Quillaja saponin (QS)-21 Solution adjuvant (QS-21), wherein the OSU-2131 doses are 80, 240 and 480 mcg in healthy volunteers and similar safety profile of the identified maximum tolerated dose (MTD) in patients awaiting solid organ transplantation.

SECONDARY OBJECTIVES:

I. Determine the optimal immunologic dose (OID) to OSU-2131 vaccination (with QS-21) in all dose cohorts of 80, 240, and 480 mcg OSU-2131 (healthy volunteers) and, upon completing safety assessment, patients awaiting solid organ transplant (PASOT).

II. To perform laboratory correlative studies to examine immune responses to the OSU-2131 vaccine with the intent to communicate the research results and to generate a de-identified data set that can then be used for future comparisons with immune response data generated in future vaccine trials.

OUTLINE: This is a dose-escalation study of OSU-2131 with fixed-dose QS-21 followed by a dose-expansion study. Healthy volunteers are randomized to 1 of 2 groups. Patients awaiting a solid organ transplant are assigned to Group I.

GROUP I (OSU-2131 WITH QS-21): Healthy volunteers and patients receive OSU-2131 subcutaneously (SC) with QS-21 SC on day 0, and weeks 2 and 4 in the absence of unacceptable toxicity or patient proceeds to transplant. Healthy volunteers and patients additionally undergo blood sample collection throughout the study.

GROUP II (PLACEBO): Healthy volunteers receive Dulbecco's phosphate-buffered saline (phosphate buffered saline [PBS]) SC on day 0, and weeks 2 and 4 in the absence of unacceptable toxicity. Healthy volunteers additionally undergo blood sample collection throughout the study.

After completion of study intervention, healthy volunteers and patients are followed up at days 29 and 35 and then at 6, 16, 28, 40 and 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and patients awaiting solid organ transplantation (SOT) must have at least one allele for HLA-B*08:01
* Subjects can be Epstein-Barr virus (EBV) seronegative or seropositive
* Subjects must be seronegative for HIV
* Subjects must be seronegative for hepatitis B and C
* Have baseline chemistry and hematology (hemoglobin, white blood cells, absolute neutrophil count, eosinophils) within normal limits
* Prothrombin time (PT) and partial thromboplastin time (PTT) below the upper limit of normal
* Platelets above the lower limit of normal (LLN)
* Basophils, lymphocytes, and monocytes must be within 1.2 x upper limit of normal (ULN) or 0.8 x LLN and considered not clinically significant by the investigator
* Total creatine kinase (CK) laboratory values < 1.25 x the upper limit of normal (according to the normal reference ranges of the Ohio State University [OSU] laboratory) at baseline (screening & pre-study visit) and considered not clinically significant by the investigator
* Subjects must not be taking antiviral therapy
* Must be ≥ 18 years of age and ≤ 65 years of age and willing to either use an effective method of contraception or abstain from sexual activity for at least 3 months following the last dose of vaccination
* Female of childbearing potential must have a negative serum pregnancy test prior to the first study drug/placebo (PBS) administration
* Agree not to receive any other investigational drug while enrolled in this study
* Provide written informed consent according to International Conference on Harmonization-Good Clinical Practice (ICH-GCP) and local regulations
* Following successful completion of safety evaluation for the phase 1 dose escalation phase of this trial in healthy volunteers and review of this data by the Sponsor and Food and Drug Administration (FDA), we plan to enroll a second cohort of patients awaiting solid organ transplantation (SOT). We will recruit patients with end stage renal disease (ESRD) who are awaiting kidney transplantation. ESRD is defined according to 2012 Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guidelines for the Evaluation and Management of Chronic Kidney Disease (Acosta-Ochoa et al, J Clin Med, 8(9):1323, 2019). KDIGO defines ESRD as: stage 4: severe reduction in glomerular filtration rate (GFR) (15 to 29 mL/min); stage 5: renal failure (GFR less than 15 mL/min). Patients will qualify for ESRD / kidney transplantation per need for maintenance dialysis due to one or more of the criteria related to renal insufficiency: volume overload, metabolic acidosis, electrolyte disturbance, drug toxicity, etc. Patients will be regularly undergoing hemodialysis or peritoneal dialysis for metabolic support. Patients will be excluded from the study if they have any unstable medical conditions which the investigator believes would preclude participation in the study. These conditions include but are not limited to cardiorenal and hepatorenal syndromes

Exclusion Criteria:

* Severe active infection, compromised cardiopulmonary function, or other serious medical illness that, in the opinion of the principal investigator, would prevent study completion
* History of chronic active EBV infection, active infectious mononucleosis (or infectious mononucleosis within 6 months of enrollment), or other EBV-related disorder as determined by principal investigator (PI)
* History of immune suppression or autoimmune disorder
* Concomitant use of systemic corticosteroids or other immunosuppressive medications (including nasal and inhaled steroids). The use of nasal steroids for seasonal rhinitis is acceptable
* Pregnant or breastfeeding subjects
* For patient enrollment on the second cohort, "patients awaiting SOT", we will consider patients awaiting kidney transplantation who are receiving maintenance renal replacement therapy (dialysis). Most patients on routine renal replacement therapy (dialysis) will present with stable chemistry, acid base balance, volume status and clear mental status. For patients who are non-compliant with routine dialysis, laboratory abnormalities and acid base, volume status can become abnormal. Specific dose limiting toxicity (DLT) criteria that may relate to patients with ESRD include laboratory parameters that may altered due to missed dialysis session(s). Most laboratory abnormalities in such patients can be corrected by restarting dialysis or blood transfusions. Outside these specific variables, we do not expect to see specific DLT criteria for patients with ESRD on this study. Metabolic derangement such as acid base imbalance, hyperkalemia and volume overload as a result of missing dialysis session. Study stopping rule for subjects awaiting organ transplant: Occurrence of this event in two or more subjects should result in study pause. Patients who are unable to adhere to routine dialysis will be excluded from the study if they have any unstable medical conditions which the investigator believes would preclude participation in the study. These conditions include but are not limited to cardiorenal and hepatorenal syndromes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From the first administration of treatment until the week 28 visit
  Will be coded to body systems and preferred terms using the Medical Dictionary for Regulatory Activities. Descriptive statistics, per treatment arm, will contain the number and percentage of subjects who experience at least one adverse event (AE), AE related to study treatment, serious AE, serious AE related to study treatment, grade 3 or 4 AE, and grade 3 or 4 related to study treatment. The number and percentage of subjects who discontinue treatment due to an AE will be provided, together with the number and percentage of subjects who die due to an AE.
Changes in laboratory parameters and vital signs | At baseline and up to week 56
  Changes will be summarized for subjects in each treatment arm. Baseline laboratory values will be summarized. The number and percentage of subjects with values below, within, and above normal range for each lab parameter will be summarized. Clinically significant abnormalities noted by the clinician during laboratory evaluations will be summarized by treatment arm.
Pre- and post-injection vital signs | Up to week 4
  The number and percent of subjects who experience a clinically significant change in vitals from pre-injection to post-injection will be tabulated and summarized by treatment arm.
Injection site reactions | At 10 and/or 60 minutes post injection on weeks 0, 2 and 4
  The number and percent of subjects who experience induration at 10 minutes post injection and/or 60 minutes post injection will be tabulated and summarized by treatment arm. The number and percent of subjects who experience erythema at 10 minutes post injection and/or 60 minutes post injection will be tabulated and summarized by treatment arm.

SECONDARY OUTCOMES:
Immune response | At baseline, day 0, and weeks 2, 4, 6, 12, 28, 40, and 56
  Will be defined as the change in pentamer RAK (RAKFKQLL) positive cells. The geometric mean of pentamer RAK positive cells will be reported at each time point with 95% confidence intervals, and the level of pentamer RAK positive cells will be plotted over time for each patient to visually identify changes in values from baseline through follow-up visits. BZLF1 HLA-B*08:01 RAK pentamers and cytometry by time-of-flight will be used to test for an immune response.
Optimal immunologic dose (OID) | Up to week 12
  Percent CD3+, CD8+, RAK+ will be quantified for each patient. This will be completed for each dose level and following dose level 3 data analysis, a collective review of the flow cytometry will be performed to aid in determining the OID.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Voorhees, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu